CLINICAL TRIAL: NCT07075939
Title: Centralization and Oncologic Outcomes in Ovarian Cancer: A Multicenter Retrospective and Prospective Observational Study Within the REMO Network (COOC-REMO)
Brief Title: Centralization and Oncologic Outcomes in Ovarian Cancer
Acronym: COOC - REMO
Status: Active, not recruiting | Type: Observational
Sponsor: Azienda USL Reggio Emilia - IRCCS (Other Government)
Collaborators: AUSL di Modena - Ospedale Ramazzini di Carpi (Unknown); AUSL di Modena - Ospedale di Mirandola (Unknown); AUSL di Modena - Ospedale Civile di Sassuolo (Unknown); AUSL di Modena - Ospedale di Pavullo nel Frignano (Unknown); AUSL di Modena - Ospedale di Vignola (Unknown); Azienda Ospedaliero-Universitaria di Modena (Other)
Responsible Party: Sponsor
Other Study IDs: 247/2025/OSS/AUSLRE
Record Dates: First submitted 2025-07-11; First posted 2025-07-20 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-07

CONDITIONS: Epithelial Ovarian Cancer; Ovarian Neoplasms; Advanced Ovarian Cancer
Keywords: ovarian cancer; Centralization of Care; COVID-19 Pandemic; Surgical Outcomes; Epithelial Ovarian Neoplasms; Progression-Free Survival; Overall Survival; Health Services Reorganization
MeSH Terms: conditions — Carcinoma, Ovarian Epithelial; Ovarian Neoplasms; COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Pre-pandemic cohort (Group A): Patients with epithelial ovarian cancer treated between January 2018 and December 2019, before the implementation of centralization policies and before the onset of the COVID-19 pandemic. Standard care was provided based on local resources and clinical practice guidelines at the time.
  Interventions: Other: No Intervention: Observational Cohort
- Pandemic peak cohort(Group B): Patients treated between January 2020 and December 2021, during the most critical phase of the COVID-19 pandemic. Centralization of care and multidisciplinary decision-making were consistently applied.Treatment decisions were influenced by reduced hospital resources, increased use of neoadjuvant chemotherapy, and enhanced centralization of surgical procedures.
  Interventions: Other: No Intervention: Observational Cohort
- Post-peak pandemic cohort(Group C): Patients treated between January 2022 and December 2023, during the phase of pandemic control. Centralization of care and multidisciplinary decision-making were consistently applied. This group reflects the new post-pandemic organizational standards.
  Interventions: Other: No Intervention: Observational Cohort

INTERVENTIONS:
Other: No Intervention: Observational Cohort — Observational data collection only

SUMMARY:
This is a multicenter, observational, retrospective and prospective study conducted within the REMO (Reggio Emilia - Modena) network in the Emilia-Romagna region (Italy), promoted by AUSL-IRCCS of Reggio Emilia.

The study aims to evaluate the impact of surgical centralization and treatment strategies adopted during the COVID-19 pandemic on oncologic outcomes in patients diagnosed with the epithelial ovarian cancer (EOC) from 2018 to 2023.

The retrospective component includes patients treated between 2018 and 2023, while the prospective component consists of clinical follow-up of those patients over the next five years.

DETAILED DESCRIPTION:
Epithelial ovarian cancer (EOC) is a highly aggressive malignancy, frequently diagnosed at an advanced stage and requiring a combined approach of surgery and systemic therapy. Complete cytoreductive surgery remains the most important prognostic factor, as residual disease ≥1 cm significantly worsens survival. In November 2019, a regional decree in Emilia-Romagna (Italy) introduced the centralization of EOC treatment to high-volume centers to improve care quality and clinical outcomes.

Shortly thereafter, the onset of the COVID-19 pandemic led to a severe reduction in healthcare resources, including surgical capacity, ICU beds, and staff availability. This situation resulted in a higher proportion of patients being referred for neoadjuvant chemotherapy, with surgery performed mainly in selected patients with better performance status and higher chances of complete resection. During this period, an increase in centralized treatments, multidisciplinary evaluations, BRCA testing, and use of interval debulking surgery (IDS) was observed.

This observational, retrospective study is designed to evaluate whether centralization and pandemic-related treatment modifications influenced oncological outcomes. The primary objective is to compare progression-free survival (PFS) and overall survival (OS) among patients treated during three different timeframes: pre-centralization/pre-pandemic (2018-2019), peak pandemic phase (2020-2021), and pandemic control phase (2022-2023). Secondary objectives include describing treatment strategies after initial diagnosis (type of surgery, chemotherapy, maintenance therapies), tumor characteristics (histology, BRCA/HRD status), recurrence patterns (site, symptoms, treatment), and the proportion of patients receiving secondary surgery, radiotherapy, Bevacizumab, and/or PARP inhibitors. No experimental interventions are included, and all patients received treatment according to routine clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Female patients aged between 18 and 99 years
* Histological and/or cytological diagnosis of epithelial ovarian cancer
* Patients evaluated by the Multidisciplinary Tumor Board (MTB) of the AUSL-IRCCS of Reggio Emilia
* Patients treated between January 1, 2018, and December 31, 2023
* Availability of clinical records and outcome data
* Signed informed consent where possible, in accordance with GDPR and Italian regulations

Exclusion Criteria:

* Patients without histological or cytological confirmation of epithelial ovarian cancer
* Incomplete or missing data for key clinical indicators
* Patients unable to provide informed consent and for whom recontact is not possible
* Patients deemed unable to understand and provide consent (e.g., severe cognitive impairment)

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Women diagnosed with epithelial ovarian cancer between January 2018 and December 2023, treated in the REMO oncological network (Reggio Emilia and Modena, Italy). Patients will be identified through retrospective review of clinical records and prospective follow-up data.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-06-27 (Actual); Primary Completion 2030-06 (Estimated); Study Completion 2030-06 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) | Up to 5 years from diagnosis
  Time from initial diagnosis of epithelial ovarian cancer to the date of first documented disease progression or death from any cause, whichever occurs first.
Overall Survival (OS) | Up to 5 years from diagnosis
  Time from initial diagnosis to death from any cause. Patients still alive will be censored at the date of last follow-up.

SECONDARY OUTCOMES:
Type of treatment received after initial diagnosis | Within 12 months from diagnosis
  Classification of treatment pathways including type of surgery (primary or interval debulking), type of chemotherapy (neoadjuvant, adjuvant, or palliative), and use of maintenance therapies.
Use of targeted therapies (Bevacizumab and/or PARP inhibitors) | Within 12 months from completion of first-line chemotherapy
  Percentage of patients treated with Bevacizumab, PARP inhibitors, or both, in adjuvant or maintenance settings.
Rate and characteristics of recurrence | Up to 5 years from diagnosis
  Frequency, site, and symptoms of disease recurrence, and rate of patients undergoing secondary surgery or radiotherapy.
Rate of radiotherapy use in recurrent disease | Up to 5 years from diagnosis
  Proportion of patients with recurrence treated with radiotherapy, including treatment site, dose, and clinical response.

CONTACTS AND LOCATIONS:
Overall Officials: Vincenzo Dario Mandato, MD, Principal Investigator — Azienda USL - IRCCS di Reggio Emilia
Locations (7):
- Italy (7):
  - Azienda Unità - Sanitaria locale di Modena - Ospedale Razzini Carpi, Carpi, Modena
  - Azienda Unità - Sanitaria locale di Modena - Ospedale di Mirandola, Mirandola, Modena
  - Azienda Unità - Sanitaria locale di Modena - Ospedale Pavullo nel Frignano, Pavullo nel Frignano, Modena
  - Azienda Unità - Sanitaria locale di Modena - Ospedale Civile Sassuolo, Sassuolo, Modena
  - Azienda Unità - Sanitaria locale di Modena - Ospedale di Vignola, Vignola, Modena
  - Azienda USL IRCCS di Reggio Emilia, Reggio Emilia, RE
  - Azienda Ospedaliero - Universitario di Modena, Modena

REFERENCES:
- [Background] Chi DS, Musa F, Dao F, Zivanovic O, Sonoda Y, Leitao MM, Levine DA, Gardner GJ, Abu-Rustum NR, Barakat RR. An analysis of patients with bulky advanced stage ovarian, tubal, and peritoneal carcinoma treated with primary debulking surgery (PDS) during an identical time period as the randomized EORTC-NCIC trial of PDS vs neoadjuvant chemotherapy (NACT). Gynecol Oncol. 2012 Jan;124(1):10-4. doi: 10.1016/j.ygyno.2011.08.014. Epub 2011 Sep 13. PMID 21917306
- [Background] Colombo N, Sessa C, Bois AD, Ledermann J, McCluggage WG, McNeish I, Morice P, Pignata S, Ray-Coquard I, Vergote I, Baert T, Belaroussi I, Dashora A, Olbrecht S, Planchamp F, Querleu D; ESMO-ESGO Ovarian Cancer Consensus Conference Working Group. ESMO-ESGO consensus conference recommendations on ovarian cancer: pathology and molecular biology, early and advanced stages, borderline tumours and recurrent disease. Int J Gynecol Cancer. 2019 May 7;29(4):728-760. doi: 10.1136/ijgc-2019-000308. PMID 31048403
- [Background] Sung H, Ferlay J, Siegel RL, Laversanne M, Soerjomataram I, Jemal A, Bray F. Global Cancer Statistics 2020: GLOBOCAN Estimates of Incidence and Mortality Worldwide for 36 Cancers in 185 Countries. CA Cancer J Clin. 2021 May;71(3):209-249. doi: 10.3322/caac.21660. Epub 2021 Feb 4. PMID 33538338
- [Background] Fotopoulou C, Concin N, Planchamp F, Morice P, Vergote I, du Bois A, Querleu D. Quality indicators for advanced ovarian cancer surgery from the European Society of Gynaecological Oncology (ESGO): 2020 update. Int J Gynecol Cancer. 2020 Apr;30(4):436-440. doi: 10.1136/ijgc-2020-001248. Epub 2020 Feb 20. No abstract available. PMID 32086362
- [Background] Goenka L, Anandaradje A, Nakka T, Kayal S, Dubashi B, Chaturvedula L, Veena P, Durairaj J, Penumadu P, Ganesan P. The "collateral damage" of the war on COVID-19: impact of the pandemic on the care of epithelial ovarian cancer. Med Oncol. 2021 Sep 28;38(11):137. doi: 10.1007/s12032-021-01588-6. PMID 34581889
- [Background] Hudry D, Becourt S, Scambia G, Fagotti A. Primary or Interval Debulking Surgery in Advanced Ovarian Cancer: a Personalized Decision-a Literature Review. Curr Oncol Rep. 2022 Dec;24(12):1661-1668. doi: 10.1007/s11912-022-01318-9. Epub 2022 Aug 15. PMID 35969358
- [Background] Mandato VD, Abrate M, De Iaco P, Pirillo D, Ciarlini G, Leoni M, Comerci G, Ventura A, Lenzi B, Amadori A, Rosati F, Martinello R, De Palma R, Ventura C, Belotti LM, Formisano D, La Sala GB; Gynecological Oncology Network of Emilia Romagna Region. Clinical governance network for clinical audit to improve quality in epithelial ovarian cancer management. J Ovarian Res. 2013 Mar 31;6(1):19. doi: 10.1186/1757-2215-6-19. PMID 23547941
- [Background] Mandato VD, Torricelli F, Uccella S, Pirillo D, Ciarlini G, Ruffo G, Annunziata G, Manzotti G, Pignata S, Aguzzoli L. An Italian National Survey on Ovarian Cancer Treatment at first diagnosis. There's None so Deaf as those who will not Hear. J Cancer. 2021 May 27;12(15):4443-4454. doi: 10.7150/jca.57894. eCollection 2021. PMID 34149908
- [Background] Mandato VD, Aguzzoli L. Management of ovarian cancer during the COVID-19 pandemic. Int J Gynaecol Obstet. 2020 Jun;149(3):382-383. doi: 10.1002/ijgo.13167. Epub 2020 Apr 29. PMID 32275775
- [Background] Mandato VD, Torricelli F, Mastrofilippo V, Pellegri C, Cerullo L, Annunziata G, Ciarlini G, Pirillo D, Generali M, D'Ippolito G, Leone C, Bologna A, Gasparini E, Palicelli A, Gelli MC, Silvotti M, Aguzzoli L. Impact of 2 years of COVID-19 pandemic on ovarian cancer treatment in IRCCS-AUSL of Reggio Emilia. Int J Gynaecol Obstet. 2023 Nov;163(2):679-688. doi: 10.1002/ijgo.14937. Epub 2023 Jun 26. PMID 37358270